CLINICAL TRIAL: NCT06503913
Title: Cognitive Muscular Therapy for Patients With Long-COVID (Post COVID-19) and Breathing Pattern Disorder
Brief Title: Cognitive Muscular Therapy for Patients With Long-COVID and Breathing Pattern Disorder
Acronym: COMLOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0186
Record Dates: First submitted 2024-07-15; First posted 2024-07-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Long COVID; Respiratory Disease
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Respiration Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Each participant will receive seven weekly sessions of Cognitive Muscular Therapy (CMT) + Breathing Visualisation at the University of Salford from an respiratory physiotherapist. This physiotherapist will have been trained to deliver the CMT intervention and will have at least three years' experience of working with patients with respiratory disorders. Each treatment session will last 45-60 mins. The CMT intervention comprises five components: Understanding long-COVID, general relaxation, postural deconstruction, contextual triggers and functional integration. Breathing Visualisation will be integrated into session 5, 6 and 7.
  Interventions: Behavioral: Cognitive Muscular Therapy; Behavioral: Breathing visualisation

INTERVENTIONS:
Behavioral: Cognitive Muscular Therapy — Psychologically informed physiotherapy which integrates training to reduce overactivity of postural muscles which can interfere with the mechanics of breathing.
Behavioral: Breathing visualisation — Breathing visualisation; Data from two 3D camera are combined and used to calculate respiratory volumes. These volumes are then used to drive an animation of breathing so that the patient can understand how their breathing pattern compares to an optimal pattern. Note this is not a medical device as data from this system is only used for education and not for diagnostic or treatment decisions.

SUMMARY:
The aim of the study is to test a treatment known as "Cognitive Muscular Therapy (CMT)" for reducing breathlessness and improving autonomic function in patients with long-COVID.

DETAILED DESCRIPTION:
A key symptom of long-COVID is dysfunctional breathing, characterised by an alteration in the muscular and mechanical control of breathing, such as altered movement/coordination of diaphragm and ribs. Long-COVID patients also experience symptoms such as dizziness and fatigue, which have been linked to dysautonomia (dysfunction of the nervous system controlling automatic body functions). Importantly, dysautonomia is connected to alterations in breathing mechanics. Specifically, rapid breathing, high in the chest, is associated with increased activity in the fight-or-flight system and decreased activity in the rest-and-repair system. Given this link, interventions capable of improving breathing mechanics could alleviate many long-COVID symptoms. However, current breathing retraining methods lack visualisation of breathing mechanics and do not integrate a whole-body approach to improving postural control.

We have developed a clinical system which can visualise breathing mechanics in real-time, providing patients with a "window into their body". We propose to integrate this system within a new intervention, known as Cognitive Muscular Therapy (CMT). CMT integrates psychological informed physiotherapy with training to reduce overactivation of postural muscles which can interfere with the mechanics of breathing. We propose to test this combined intervention on 20 people with Long-COVD to understand if we can improve respiratory function and symptoms associated with dysautonomia. If successful, this pilot study could pave the way for large-scale studies in long-COVID

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Experience moderate/severe breathlessness, quantified using the Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) scale.
* Speak and understand English sufficiently to read the information sheet and sign the consent form
* Ability to stand without any assistive device for at least 20 minutes (to ensure sufficient capacity to complete the intervention)

Exclusion Criteria:

* Dementia or other major cognitive impairment
* BMI >32 (as increased subcutaneous fat prevents use of breathing measurement system)
* Current smoker or smoked regularly within last 6 months
* Any cardiorespiratory disease that requires medical intervention (except asthma management)
* Currently receiving physiotherapy-based treatment for LC or breathing pattern disorder
* Significant respiratory co-morbidity (e.g. COPD, uncontrolled Asthma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Nijmegen Questionnaire | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture breathlessness symptoms associated with hyperventilation disorder. Score 0 - 60 (0 = no hyperventilation symptoms, 60 severe symptoms of hyperventilation).

SECONDARY OUTCOMES:
Change in Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) scale | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture breathlessness symptoms associated with long-COVID compared to pre-acute infection. Score 0 - 45 (0 = no long-COVID symptoms, 45 severe symptoms of long-COVID).
Change in Dyspnea-12 questionnaire | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture breathlessness symptoms. Score 0 - 36 (0 = no breathlessness symptoms, 36 severe breathlessness).
Change in Self-evaluation of breathing questionnaire | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture breathlessness symptoms associated with dysfunctional breathing. Score 0 - 75 (0 = no dysfunctional breathing symptoms, 60 severe symptoms of dysfunctional breathing).
Change in Composite Autonomic Symptom Score | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture symptoms associated with autonomic dysfunction. 31 questions rating the symptoms associated with autonomic dysfunction.
Change in EQ-5D-5L | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture an individual's quality of life through their ability to complete daily living activities. Each heading is rated from no problems through to unable to complete the task.
Change in WHO Disability Assessment Schedule (12-item) | Change from Baseline to two months (post intervention) & change from Baseline to 5 months (post intervention)
  Used to capture an individual's ability to perform daily living activities. Each point is rated from No difficulty performing a task to extreme difficulty/cannot complete the task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no data sharing plan